CLINICAL TRIAL: NCT07240740
Title: WittyChildren: a Quantitative Evaluation of Motor-cognitive Coordination
Brief Title: WittyChildren - Advanced Technology for Response Time Evaluation in Children Affected by Developmental Disorders
Status: Completed | Type: Observational
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Sponsor
Other Study IDs: 984
Record Dates: First submitted 2025-04-30; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: The WittySEM system, in addition to simultaneously allowing the evaluation of the movement associated with the execution of the task, also provides for an active and "play-like" involvement of the sub — The possibility of using tools for objective and quantitative evaluations can overcome these limitations. Added to this is the need to evaluate the beneficial effects of rehabilitation so as to understand its effectiveness and impact on quality of life. However, it is difficult to resort to tests that use dedicated devices such as the WittySEM system which, in addition to simultaneously allowing the evaluation of the movement associated with the execution of the task, also provides for an active and "play-like" involvement of the subject which should not be underestimated in the case of children.

SUMMARY:
The WittyChildren project aims to evaluate the response to visual stimuli in terms of reaction times and movement execution using advanced instruments. The evaluation is aimed at children with motor and cognitive deficits associated with various pathologies such as Down Syndrome, Infantile Cerebral Palsy, Autism. The evaluation protocol involves the execution of specific memory tasks: the child is asked to turn off light targets equipped with proximity sensors by approaching their hand. These visual signals, consisting of colored lights and symbols, are emitted according to pre-established patterns by a dedicated LED system (WittySEM - Microgate) capable of precisely measuring reaction times. During the execution of the task, quantitative and multifactorial analysis of movement and posture is also performed using an optoelectronic system (Smart DX - BTS Bioengineering) in order to obtain a complete analysis obtained from the combination of information regarding the child's motor and cognitive abilities. The analysis is repeated pre- and post-specific rehabilitation treatment, such as ARMEO, CIMT and occupational therapy, with the aim of evaluating the effects with objective and quantitative measurements through cutting-edge instruments, thus overcoming the intrinsic limits of commonly used scales and clinical tests. The project will be implemented in collaboration with the Politecnico di Milano - Lecco Territorial Campus and the IRCCS Eugenio Medea - Associazione la nostra famiglia. The first will provide the study with the necessary equipment at the "Human Performance Laboratory - E4Sport" of the Lecco Territorial Campus and the biomechanical engineering skills. The second, thanks to its consolidated experience in the treatment, rehabilitation and research of childhood pathologies, will provide the necessary support from a medical/rehabilitative point of view.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric age (< 18 years);
* Diagnosis of hemiplegia or hemiplegic CP;
* Ability to understand and follow given motor instructions;
* Ability to move such that the use of crutches or wheelchairs is not required.

Exclusion Criteria:

* Severe cognitive impairment.
* Severe visual impairment
* Uncontrolled epilepsy

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients affected by unilateral cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Reaction time - before rehabilitation | Baseline, before starting rehabilitation treatment
  Reaction time as measured through optoelectronic data.
Reaction time - after rehabilitation | After one month
  Reaction time as measured through optoelectronic data.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS E. Medea, Bosisio Parini, LC, Italy